CLINICAL TRIAL: NCT00924248
Title: Primovist Regulatory Post Marketing Surveillance
Brief Title: Primovist Regulatory Post Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare AG
Other Study IDs: 14332; PR0810KR (Other: company internal)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Liver
Keywords: Liver MRI
MeSH Terms: interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Gadoxetic acid disodium (Primovist, BAY86-4873)

INTERVENTIONS:
Drug: Gadoxetic acid disodium (Primovist, BAY86-4873) — Patients in daily life clinical practice treatment receiving Primovist according to indication on the label.

SUMMARY:
The objective of this Post Marketing Surveillance (PMS) is to gain information about safety and efficacy in real practice

ELIGIBILITY:
Inclusion Criteria:

* Patient who take Primovist for liver MRI

Exclusion Criteria:

* Patients who belong to the contraindication on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean who take Primovist for liver MRI
Sampling Method: Non-Probability Sample
Enrollment: 4358 (Actual)
Dates: Start 2007-10; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety evaluation in real practice (SAE/AE/ADR collection) | After administration

SECONDARY OUTCOMES:
Assessment of contrast effect by imaging after administration | Before administration
Overall contrast effects by combining individual assessment | Before administration
Assessment of contrast enhancement effect | After administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea